CLINICAL TRIAL: NCT03011593
Title: Effect of UGIR on Quality of Life in Adults With Compromised Gut Function and Malabsorption
Brief Title: Effect of UGIR in Adults With Compromised Gut Function and Malabsorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metagenics, Inc. (Industry)
Collaborators: National University of Natural Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UGIR
Record Dates: First submitted 2016-12-14; First posted 2017-01-05 (Estimated); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Irritable Bowel Syndrome; Crohn Disease; Ulcerative Colitis; Celiac Disease
MeSH Terms: conditions — Irritable Bowel Syndrome; Crohn Disease; Colitis, Ulcerative; Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nutrition Support Product (Experimental): Participants were asked to take a nutrition support product twice per day for a period of 6 weeks.
  Interventions: Other: Nutrition Support Product

INTERVENTIONS:
Other: Nutrition Support Product — Nutrition support product contains macronutrients, micronutrients, glutamine, and prebiotics. Product is in powder form (41 grams per serving) and is mixed with water or juice before consumption. Taken orally as a nutritional shake twice per day.
  Other Names: UGIR

SUMMARY:
This study assessed the effect of a nutrition support product on quality of life in adults with compromised gut function and malabsorption.

DETAILED DESCRIPTION:
This prospective, non-randomized, open-label study assessed the effect of a nutrition support product on quality of life in adults with compromised gut function and malabsorption. Adults with irritable bowel syndrome (IBS), inflammatory bowel disease (IBD) or celiac disease were enrolled in the study and asked to take the study product for 6 weeks. The primary measure of the study was a validated quality of life questionnaire, the Gastrointestinal Quality of Life Index (GIQLI). Secondary measures included the Inflammatory Bowel Disease Questionnaire (IBDQ), the Celiac Disease Questionnaire (CDQ), and the Digestive Symptom Frequency Questionnaire (DSFQ).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 19 - 40 kg/m2
* Previous diagnosis of ulcerative colitis (UC), Crohn's disease, irritable bowel syndrome (IBS), or celiac disease

Exclusion Criteria:

* Gastroenterologic surgery within 3 months before the study period
* Have a colostomy or ileostomy bag
* Malignancy within the last 5 years
* Women who are lactating, pregnant or planning pregnancy during the study period
* Taking antibiotic, antiparasitic, or antifungal medications
* Initiation of or changes to supplements or medications within 28 days prior to screening

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Gastrointestinal Quality of Life Index (GIQLI) Score | 6 weeks

SECONDARY OUTCOMES:
Change in Inflammatory Bowel Disease Questionnaire (IBDQ) Score | 6 weeks
Change in Celiac Disease Questionnaire (CDQ) Score | 6 weeks
Change in Digestive Symptom Frequency Questionnaire (DSFQ) Score | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nikhat Contractor, PhD, Study Director — Metagenics, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ryan JJ, Monteagudo-Mera A, Contractor N, Gibson GR. Impact of 2'-Fucosyllactose on Gut Microbiota Composition in Adults with Chronic Gastrointestinal Conditions: Batch Culture Fermentation Model and Pilot Clinical Trial Findings. Nutrients. 2021 Mar 14;13(3):938. doi: 10.3390/nu13030938. PMID 33799455
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33799455/